CLINICAL TRIAL: NCT03665961
Title: The Association Between Microbiota, Endotoxaemia and the Host Obesity/ Insulin Resistance (MiPOOP Study)
Acronym: MiPOOP
Status: Completed | Type: Observational
Sponsor: Changi General Hospital (Other)
Collaborators: Genome Institute of Singapore (Other)
Responsible Party: Principal Investigator, John Chen Hsiang, Consultant, Changi General Hospital
Other Study IDs: MiPOOP
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Central Obesity
Keywords: gastrointestinal microbiome; metabolic syndrome; ethnicity; dietary components
MeSH Terms: conditions — Obesity, Abdominal; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Microbial DNA from stool samples, genomic DNA from whole blood, and plasma samples from whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central obesity: Cases with central obesity as defined by waist circumference cut-offs ≥ 90 cm in men and ≥ 80 cm in women for Asians
- No central obesity: Controls with no central obesity

SUMMARY:
The objectives of this study are to examine the effects of ethnicity, central obesity and dietary components, on the human gut microbiome. The investigators hypothesize that these factors have an influence on the composition of the gut microbiome. Healthy subjects (n=35) provided stool samples for gut microbiome profiling using 16S rRNA sequencing and completed a dietary questionnaire. The serum samples were assayed for a panel of inflammatory cytokines. Their associations with central obesity were examined.

DETAILED DESCRIPTION:
Introduction: Perturbance in the composition of human gut microbiota has been associated with metabolic disorders such as obesity, diabetes mellitus and insulin resistance. The objectives of this study are to examine the effects of ethnicity, central obesity and dietary components, on the human gut microbiome. The investigators hypothesize that these factors have an influence on the composition of the gut microbiome.

Methods: Subjects of Chinese (n=14), Malay (n=10) or Indian (n=11) ancestry, median age 39 (range:22-70 years old), were enrolled. The subjects provided stool samples for gut microbiome profiling using 16S rRNA sequencing and completed a dietary questionnaire. The serum samples were assayed for a panel of biomarkers (Interleukin-6, tumour necrosis factor alpha, adiponectin, cleaved cytokeratin 18, lipopolysaccharide binding protein and limulus amebocyte lysate). Central obesity was defined by waist circumference cut-offs in Asians.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent,
* Aged between 21- 75 years old,
* Body Mass Index (BMI) of > 18 kg/m2,
* Ethnic group of either Chinese, Malay or Indian as evidenced by identification card,
* Subject with absence of impaired glucose tolerance,
* Subject is healthy with no clinically significant disease or condition as determined through their medical history, physical examination; Diabetes mellitus was defined as Type 2 DM fulfilling the WHO criteria and the care of Department of Endocrinology, Changi General Hospital,
* Ability to communicate with investigator and to understand and comply with all requirements of study participation.

Exclusion Criteria:

* Subject who are viral Hepatitis (B or C) or HIV positive as per declaration,
* Subject who had bariatric surgery including lap banding, gastric sleeve surgery, cholecystectomy,
* Subject who has > 5% weight loss in the last 3 months prior to study enrolment as per declaration,
* Subject who are on 'stable' insulin sensitizers such as such as rosiglitazone, metformin for the last 3 months prior to enrolment,
* Pregnant women,
* Subject who has been treated with antibiotics within 6 weeks of enrolment,
* Subject who has usage of lactulose, dietary fibres for purpose of constipation,
* Subject with immune-compromised status; undergoing chemotherapy, on steroid,
* Subject with FMHx or PMHx of autoimmune disease, GI cancers, inflammatory bowel disease, Irritable bowel syndrome and anxiety or depression as per declaration.

Ages: 21 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers recruited through advertisement or patients with type 2 diabetes mellitus from hospital records.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Association of human gut microbiome profile with central obesity and dietary pattern | 1 day
  Species diversity as measured by diversity indices

SECONDARY OUTCOMES:
Association of human gut microbiome profile with ethnicity | 1 day
  Species diversity as measured by diversity indices
Association of interleukin-6 with central obesity and microbiota | 1 day
  Interleukin-6 concentration in pg/ml
Association of tumour necrosis factor - alpha with central obesity and microbiota | 1 day
  Tumour necrosis factor - alpha concentration in pg/ml
Association of cleaved cytokeratin 18 with central obesity and microbiota | 1 day
  Cleaved cytokeratin 18 concentration in units/L
Association of limulus amebocyte lysate with central obesity and microbiota | 1 day
  Limulus amebocyte lysate concentration in EU/ml
Association of lipopolysaccharide binding protein with central obesity and microbiota | 1 day
  Lipopolysaccharide binding protein concentration in ng/ml
Analysis of dietary components based on recommended daily allowance | 3 days
  Dietary questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: John Chen Hsiang, MD, PhD, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsiang JC, Bai WW, Raos Z, Stableforth W, Upton A, Selvaratnam S, Gane EJ, Gerred SJ. Epidemiology, disease burden and outcomes of cirrhosis in a large secondary care hospital in South Auckland, New Zealand. Intern Med J. 2015 Feb;45(2):160-9. doi: 10.1111/imj.12624. PMID 25371019
- [Background] Ho EXP, Cheung CMG, Sim S, Chu CW, Wilm A, Lin CB, Mathur R, Wong D, Chan CM, Bhagarva M, Laude A, Lim TH, Wong TY, Cheng CY, Davila S, Hibberd M. Human pharyngeal microbiota in age-related macular degeneration. PLoS One. 2018 Aug 8;13(8):e0201768. doi: 10.1371/journal.pone.0201768. eCollection 2018. PMID 30089174